CLINICAL TRIAL: NCT07169968
Title: Evaluation of the Effects of Micro-Osteoperforations on The Efficiency of Orthodontic Clear Aligner Therapy for Alleviating Mandibular Anterior Crowding: A Randomized Clinical Trial
Brief Title: Effects of Micro-osteoperforations on Lower Anterior Crowding Using Clear Aligners
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec ID052429
Record Dates: First submitted 2025-08-21; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-06

CONDITIONS: Mandibular Dental Crowding
Keywords: Micro-osteoperforations; aligner tracking; lower anterior crowding; clear aligners
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: Clear aligner treatment (Active Comparator): the control group that will receive clear aligner treatment for lower anterior treatment without micro-osteoperforations
  Interventions: Device: clear aligners group
- group 2: clear aligner treatment with micro-osteoperforations (Experimental): the experimental group that will receive clear aligner treatment for lower anterior treatment with micro-osteoperforations using mini-implants for acceleration of tooth movement and improving aligner's tracking
  Interventions: Device: micro-osteoperforations group

INTERVENTIONS:
Device: clear aligners group — patients with lower anterior crowding, after randomization and allocation, will receive intraoral scanning to create a digital model. using computer software, teeth segmentation, setup and stagging of tooth movement will be carried out. models for each stage of tooth movement will be three-dimentionally printed and the aligners will be thermoformed over each model. patients are instructed to wear each aligner for a week then continue to the next aligner till treatment is finished
  Other Names: control group; group 1
  Arms: group 1: Clear aligner treatment
Device: micro-osteoperforations group — patients having lower anteriro crowding, after randomization and allocation, aligners will be produced for them. patients in this group will receive micro-osteoperforation using mini-implants before wearing the first aligner and after one month from starting treatment.
  Other Names: experimental group; group 2
  Arms: group 2: clear aligner treatment with micro-osteoperforations

SUMMARY:
this randomized controlled trial is designed to compare between clear aligner therapy in alleviating mandibular anterior crowding alone versus with micro-osteoperforations

DETAILED DESCRIPTION:
This study is carried on in order to provide a method to enhance the predictability of clear aligner treatment. Loss of aligner tracking is one of the problems encountered during aligner treatment that results in increasing number of aligners required to complete treatment in addition to increasing the overall treatment time and cost. Micro-osteoperforation is a method for acceleration of orthodontic tooth movement and could be used to improve tooth movement and predictability of treatment with clear aligners. So this study is aimed to evaluate the efficiency of aligner treatment during alleviation of lower anterior crowding with and without micro-osteoperforations

ELIGIBILITY:
Inclusion Criteria

1. Adult patients with age ranging from 18 to 35 years.
2. Healthy periodontium.
3. Presence of full set of permanent dentition excluding third molars.
4. Patients requiring non-extraction orthodontic treatment in the mandibular arch.
5. Mandibular anterior little's irregularity index from 3 to 6.
6. No spaces in the mandibular arch.

Exclusion Criteria:

1. Presence of retained primary teeth in the mandibular arch.
2. Patients having systemic diseases as (e.g., diabetes, osteoporosis) or taking medication that could affect tooth movement (e.g., bisphosphonates, anticancer drugs)
3. Vulnerable patients.
4. Smokers.
5. Pregnant female patients.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
aligner effectivness | 3-9 months
  Number of aligners prescribed versus required (total number of aligners including refinements) for each group

SECONDARY OUTCOMES:
relief of dental crowding | 3-9 months
  relief of crowding will be assessed using Little's Irregularity Index
gingival assessment | 3-9 months
  measuring gingival index before and after treatment
pain assessment | from day 1 to day 7 after micro-osteoperforations
  evaluating pain experienced after micro-osteoperforation using Visula Analoge score (VAS)
periodontal assessment | 3-9 months
  measuring periodontal pocket depth before and after teatment
tooth mobility assessment | 3-9 months
  measuring mobility index before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of orthodontics, Faculty of Dentistry, Ain Shams University, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No